CLINICAL TRIAL: NCT06372171
Title: Effects of Liposomal Encapsulation on Vitamin C Absorption and Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, YenPing, Lei, Assistant professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NYCU112182AEF
Record Dates: First submitted 2024-03-24; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Other): Day 14
  Interventions: Dietary Supplement: Satge 1
- Stage 2 (Other): Day 28
  Interventions: Dietary Supplement: Stage 2

INTERVENTIONS:
Dietary Supplement: Satge 1 — General vitamin C powder group (Contains 1500 mg Vitamin C) Number 1-10 liposomal encapsulation C powder group (Contains 1500 mg of vitamin C and lecithin and is coated) Number 11-20
  Arms: Stage 1
Dietary Supplement: Stage 2 — General vitamin C powder group (Contains 1500 mg Vitamin C) Number 11-20 liposomal encapsulation C powder group (Contains 1500 mg of vitamin C and lecithin and is coated) Number 1-10
  Arms: Stage 2

SUMMARY:
Vitamin C is an important antioxidant in the human body and plays many important roles. It is currently known that vitamin C has the functions of treating scurvy, assisting in collagen synthesis, whitening, and increasing immunity. Smokers, patients with cardiovascular disease, and patients with diabetes may have higher requirements for vitamins due to higher oxidative stress in the body. Liposome coating is a technology commonly used in food processing and medicine to protect active substances, increase absorption or slow release. Currently, vitamin C is commonly available on the market as an additive nutritional supplement in the form of powder packets, tablets, etc. The disadvantages are that vitamin C is relatively unstable, easily destroyed by gastric acid, and maintains blood concentration for a short time. Taking liposome microbial C has been Found to have the potential to increase bioavailability in the human body, it is expected that vitamin C coated with lecithin is relatively stable and can be stabilized in the small intestine without being damaged by gastric acid, while reducing the risk of gastrointestinal discomfort caused by the acidity of vitamin C. According to the revised seventh edition of the Reference Intake of Dietary Nutrients for Chinese People, the upper daily intake of vitamin C (tolerable upper intake levels, UL) for people aged 19 to 70 is 2,000 mg. According to literature, the absorption rate of vitamin C when consuming 30-180 mg per day is about 70-90%; when the daily intake exceeds 1000 mg, the absorption rate will drop to less than 50%. The dose of vitamin C used in this study is more than 1500 mg. The purpose is to explore whether the sustained-release characteristics of liposome coating technology can improve the absorption rate and achieve better bioavailability when consuming high-dose vitamin C powder. It is expected that through the egg The liposome vitamin C powder made of phospholipids increases its maintenance time in the blood, thereby increasing the supplementary effect of vitamin C powder and serving as another supplement option for vitamin C.

DETAILED DESCRIPTION:
The trial is divided into two parts, the first part is "pre-trial screening" and the second part is "clinical trial".

This trial will first conduct the following tests to confirm that the subjects meet the inclusion and exclusion conditions before screening before they are eligible for the formal trial.

1. General examination (height, weight, blood pressure)
2. Blood biochemical index detection (fasting blood glucose, triglycerides, total cholesterol, Blood urea nitrogen, Creatinine, GOT, GPT), single blood draw volume: 3 c.c., frequency: 1 time, total blood volume: 3 c.c.

It is expected to recruit 20 eligible healthy subjects. This trial adopts a two-stage open crossover trial (Crossover) design. After the subjects join the trial, they need to participate in a total of 2 trials. After each trial is completed, a 14-day interval (washout period) is required before the next trial (the first trial) can be conducted. → 14 days apart → second test). At the beginning of the experiment, the subjects drew lots to determine their numbers and the order of participating groups (the participating groups in the two experiments will not be repeated).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-60 years old, without heart, liver, kidney, endocrine or major organic diseases (patient report), and able to fully cooperate with the experiment.

Exclusion Criteria:

1. Patients with renal insufficiency and dialysis
2. Cancer patients
3. Underweight (BMI≦17) or obese (BMI≧27)
4. Those taking medications for chronic diseases
5. Blood pressure systolic blood pressure ≧ 130 mmHg or diastolic blood pressure ≧ 85 mmHg
6. Fasting blood glucose ≧ 100 mg/dL
7. Fasting triglycerides ≧ 150 mg/dL, total cholesterol ≧ 200 mg/dL
8. Have a history of vitamin C allergy
9. People suffering from mental illness
10. Pregnant and breastfeeding women
11. Patients with hemosiderosis
12. Kidney stone patients
13. People who take vitamin C for a long time should take supplements (at least 200 mg per day for more than one month)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
General examination | Day 14 and 28
  BMI(Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared) and blood pressure
Hematology Test | Day 14 and 28
  Fasting blood glucose, triglycerides, total cholesterol, Blood urea nitrogen, Creatinine(Blood urea nitrogen (BUN) and creatinine tests can be used together to find the BUN-to-creatinine ratio (BUN:creatinine). A BUN-to-creatinine ratio can help your doctor check for problems, such as dehydration, that may cause abnormal BUN and creatinine levels.), GOT, GPT

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Beitou Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No